CLINICAL TRIAL: NCT02833363
Title: Difference of Gastric Microbiota in the Process of Correa's Model.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-08
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Microbiota; Non-atrophic Gastritis; Atrophic Gastritis; Intestinal Metaplasia; Intraepithelial Neoplasia; Gastric Cancer; Helicobacter Pylori
Keywords: gastric microbiota; Helicobacter pylori; Non-atrophic Gasrititis; Atrophic gastritis; Intestinal metaplasia; intraepithelial neoplasia; Gastric cancer
MeSH Terms: conditions — Gastritis, Atrophic; Carcinoma in Situ; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gastric mucosal samples from antrum and corpus will be collected during gastroscopy,and used for microbiota analysis by high-throughput sequencing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- patients with non-atrophic gastritis
- Patients with gastritis
- Patients with intestinal metaplasia
- Patients with intrepithelial neoplasia
- Patients with non-cardia gastric cancer

SUMMARY:
Helicobater pylori plays an important role in the development of gastric cancer. Eradication therapy can reducing the morbidity of gastric cancer, but can't totally prevent it especially when atrophy and more serious precancerous lesions already happened. Prior studies found the gastric bacterial difference among gastritis, intestinal metaplasia and gastric cancer. However, they didn't reach an agreement. Correa's model is widely accepted in the development of gastric cancer. The pathological change makes a more suitable environment for bacteria to overgrowth. This study are designed to analyze the gastric microbial difference of non-atrophic gastritis, atrophic gastritis, intestinal metaplasia, intraepithelial neoplasia and gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients go through a gastric endoscopy examination with non-atrophic gastritis, atrophic gastris, intestinal metaplasia, intraepithelial neoplasia and gastric cancer.
2. Did not take any antibiotics,PPI,probiotics and chinese herbs in the past one month,and took less than one week in the past three months before the gastroscopy examination.
3. Sign the informed consent.

Exclusion Criteria:

1. Had been taken Helicobacter pylori eradication therapy before.
2. Previous gastrointestinal surgery.
3. During the pregnancy and lactation period.
4. With any serious diseases like liver failure,heart failure,renal failure,malignant tumor,alcoholism or any other disease that may effect the result.
5. With any mental problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients go through a gastric endoscopy examination with non-atrophic gastritis, atrophic gastris, intestinal metaplasia, intraepithelial neoplasia and gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Difference of Gastric Microbiota in the Process of Correa's Model. | 5 months

SECONDARY OUTCOMES:
Difference of Gastric Microbiota in the Process of Correa's Model. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD,PHD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China